CLINICAL TRIAL: NCT01072279
Title: Strengthening and Evaluating the "Preventing Malnutrition in Children Under Two Years of Age Approach" (PM2A) in Guatemala and Burundi
Brief Title: Preventing Malnutrition in Children Under Two Years of Age Approach
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: International Food Policy Research Institute (Other)
Collaborators: Food and Nutrition Technical Assistance Project 2 of the Academy of Educational Development (Unknown); United States Agency for International Development (USAID) (U.S. Federal Agency); Catholic Relieve Services-Burundi (Unknown); Mercy Corps-Guatemala (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 4001-IFPRI-00
Record Dates: First submitted 2010-02-17; First posted 2010-02-22 (Estimated); Last update posted 2016-02-25 (Estimated); Status verified 2013-01

CONDITIONS: Malnutrition
Keywords: Malnutrition;; Infant nutrition;; Fortified food; Linear growth; Cluster randomized controlled trials; Effectiveness; Impact evaluation studies; Burundi; Guatemala
MeSH Terms: conditions — Malnutrition

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (10):
- Burundi: T24 (Experimental)
  Interventions: Other: Tubaramure (Burundi)
- Burundi: TNFP (Experimental)
  Interventions: Other: Tubaramure (Burundi)
- Burundi: T18 (Experimental)
  Interventions: Other: Tubaramure (Burundi)
- Burundi: Control (No Intervention)
- Guatemala: PROCOMIDA (Experimental)
  Interventions: Other: Procomida (Guatemala)
- Guatemala: no family ration (Experimental)
  Interventions: Other: Procomida (Guatemala)
- Guatemala: LNS (Experimental)
  Interventions: Other: Procomida (Guatemala)
- Guatemala: Sprinkles (Experimental)
  Interventions: Other: Procomida (Guatemala)
- Guatemala: reduced family ration (Experimental)
  Interventions: Other: Procomida (Guatemala)
- Guatemala: control (No Intervention)

INTERVENTIONS:
Other: Tubaramure (Burundi) — Different combinations of family food rations, individual food rations, micronutrient supplements and behavior change communication to encourage optimal and age-appropriate infant and child feeding practices
  Arms: Burundi: T18; Burundi: T24; Burundi: TNFP
Other: Procomida (Guatemala) — Different combinations of family food rations, individual food rations, micronutrient supplements and behavior change communication to encourage optimal and age-appropriate infant and child feeding practices
  Arms: Guatemala: LNS; Guatemala: PROCOMIDA; Guatemala: Sprinkles; Guatemala: no family ration; Guatemala: reduced family ration

SUMMARY:
A study conducted by IFPRI in Haiti provided the first programmatic evidence, using a cluster randomized evaluation design, that preventing child undernutrition in children under two years of age (PM2A) through an integrated program providing food rations, BCC and preventive health and nutrition services is both feasible and highly effective. The study's principal aim was to compare a newly designed preventive approach with the traditional (recuperative) food assisted MCHN program approach, and therefore included only two comparison groups: one group of communities that was randomly assigned to the preventive approach and another group assigned to the recuperative approach. For logistical and financial reasons, the study did not include a randomized control group receiving no intervention.

The Haiti study design was well-suited to achieve its main goal - i.e. to test whether the preventive approach was more effective than the recuperative approach at preventing child undernutrition - but it left a number of questions unanswered.

The present study will address several of these questions, which will allow to further refine the PM2A approach, facilitate its replication in different contexts, and maximize its impact and cost-effectiveness in future programming. The study will be conducted in Guatemala and Burundi. The key research objectives are:

1. Impact and cost effectiveness: Assess the impact and cost effectiveness of PM2A on child nutritional status.
2. Optimal composition and size of food rations in PM2A: Assess the differential and absolute impact of varying the size and types of foods incorporated in the food ration of the PM2A. More specifically, assess the differential effect of different sizes of family food rations, and assess the impact of substituting the individual food ration with new micronutrient-rich products such as lipid-based nutrient supplements (LNS) or micronutrient Sprinkles.
3. Optimal timing and duration of PM2A: Assess the differential and absolute impact of varying the timing and duration of exposure to PM2A on child nutritional status.

ELIGIBILITY:
Inclusion Criteria:

* Guatemala: pregnant mothers and subsequently their born children up to the age of 24 months;
* Burundi: cross-sectional study: children 0 to 42 of age.

Exclusion Criteria:

* none

Max Age: 42 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 16895 (Actual)
Dates: Start 2010-04; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
child nutritional status | Burundi: 2 years; Guatemala: at pregnancy, 1 mo, 4 mo, 6 mo, 9 mo, 12 mo, 18 mo, 24 mo

SECONDARY OUTCOMES:
household food security | Burundi: after 2 years; Guatemala: at pregnancy, 1 mo, 4 mo, 6 mo, 9 mo, 12 mo, 18 mo, 24 mo
household food and non-food consumption | Burundi: after 2 years; Guatemala: at pregnancy, 1 mo, 4 mo, 6 mo, 9 mo, 12 mo, 18 mo, 24 mo
maternal knowledge on infant and young child feeding (IYCF) and health | Burundi: after 2 years; Guatemala: at pregnancy, 1 mo, 4 mo, 6 mo, 9 mo, 12 mo, 18 mo, 24 mo
attitudes towards IYCF and health | Burundi: after 2 years; Guatemala: at pregnancy, 1 mo, 4 mo, 6 mo, 9 mo, 12 mo, 18 mo, 24 mo
morbidity | Burundi: after 2 years; Guatemala: at pregnancy, 1 mo, 4 mo, 6 mo, 9 mo, 12 mo, 18 mo, 24 mo
health care seeking behavior | Burundi: after 2 years; Guatemala: at pregnancy, 1 mo, 4 mo, 6 mo, 9 mo, 12 mo, 18 mo, 24 mo

CONTACTS AND LOCATIONS:
Overall Officials: Marie Ruel, PhD, Principal Investigator — IFPRI
Locations (2):
- CRS Burundi, Bujumbura, Burundi
- Guatemala: Mercy Corps, Guatemala: Coban, Guatemala

REFERENCES:
- [Background] Loechl CU, Menon P, Arimond M, Ruel MT, Pelto G, Habicht JP, Michaud L. Using programme theory to assess the feasibility of delivering micronutrient Sprinkles through a food-assisted maternal and child health and nutrition programme in rural Haiti. Matern Child Nutr. 2009 Jan;5(1):33-48. doi: 10.1111/j.1740-8709.2008.00154.x. PMID 19161543
- [Background] Menon P, Mbuya M, Habicht JP, Pelto G, Loechl CU, Ruel MT. Assessing supervisory and motivational factors in the context of a program evaluation in rural Haiti. J Nutr. 2008 Mar;138(3):634-7. doi: 10.1093/jn/138.3.634. PMID 18287379
- [Background] Ruel MT, Menon P, Habicht JP, Loechl C, Bergeron G, Pelto G, Arimond M, Maluccio J, Michaud L, Hankebo B. Age-based preventive targeting of food assistance and behaviour change and communication for reduction of childhood undernutrition in Haiti: a cluster randomised trial. Lancet. 2008 Feb 16;371(9612):588-95. doi: 10.1016/S0140-6736(08)60271-8. PMID 18280329
- [Background] Menon P, Ruel MT, Loechl CU, Arimond M, Habicht JP, Pelto G, Michaud L. Micronutrient Sprinkles reduce anemia among 9- to 24-mo-old children when delivered through an integrated health and nutrition program in rural Haiti. J Nutr. 2007 Apr;137(4):1023-30. doi: 10.1093/jn/137.4.1023. PMID 17374671
- [Background] Menon P, Ruel MT, Loechl C, Pelto G. From research to program design: use of formative research in Haiti to develop a behavior change communication program to prevent malnutrition. Food Nutr Bull. 2005 Jun;26(2):241-2. doi: 10.1177/156482650502600210. No abstract available. PMID 16060227
- [Background] Ruel MT, Menon P, Loechl C, Pelto G. Donated fortified cereal blends improve the nutrient density of traditional complementary foods in Haiti, but iron and zinc gaps remain for infants. Food Nutr Bull. 2004 Dec;25(4):361-76. doi: 10.1177/156482650402500406. PMID 15646314
- [Derived] Leroy JL, K Olney D, Bliznashka L, Ruel M. Tubaramure, a Food-Assisted Maternal and Child Health and Nutrition Program in Burundi, Increased Household Food Security and Energy and Micronutrient Consumption, and Maternal and Child Dietary Diversity: A Cluster-Randomized Controlled Trial. J Nutr. 2020 Apr 1;150(4):945-957. doi: 10.1093/jn/nxz295. PMID 31858128
- [Derived] Leroy JL, Olney DK, Ruel MT. PROCOMIDA, a Food-Assisted Maternal and Child Health and Nutrition Program, Contributes to Postpartum Weight Retention in Guatemala: A Cluster-Randomized Controlled Intervention Trial. J Nutr. 2019 Dec 1;149(12):2219-2227. doi: 10.1093/jn/nxz175. PMID 31373374
- [Derived] Olney DK, Leroy JL, Bliznashka L, Ruel MT. A Multisectoral Food-Assisted Maternal and Child Health and Nutrition Program Targeted to Women and Children in the First 1000 Days Increases Attainment of Language and Motor Milestones among Young Burundian Children. J Nutr. 2019 Oct 1;149(10):1833-1842. doi: 10.1093/jn/nxz133. PMID 31268132
- [Derived] Olney DK, Leroy J, Bliznashka L, Ruel MT. PROCOMIDA, a Food-Assisted Maternal and Child Health and Nutrition Program, Reduces Child Stunting in Guatemala: A Cluster-Randomized Controlled Intervention Trial. J Nutr. 2018 Sep 1;148(9):1493-1505. doi: 10.1093/jn/nxy138. PMID 30184223
- [Derived] Leroy JL, Olney D, Ruel M. Tubaramure, a Food-Assisted Integrated Health and Nutrition Program, Reduces Child Stunting in Burundi: A Cluster-Randomized Controlled Intervention Trial. J Nutr. 2018 Mar 1;148(3):445-452. doi: 10.1093/jn/nxx063. PMID 29546306
- [Derived] Leroy JL, Olney D, Ruel M. Tubaramure, a Food-Assisted Integrated Health and Nutrition Program in Burundi, Increases Maternal and Child Hemoglobin Concentrations and Reduces Anemia: A Theory-Based Cluster-Randomized Controlled Intervention Trial. J Nutr. 2016 Aug;146(8):1601-8. doi: 10.3945/jn.115.227462. Epub 2016 Jul 13. PMID 27412269